CLINICAL TRIAL: NCT06955481
Title: Prospective, Single-arm, Multicenter Study to Evaluate the Performance of Navigated Total Knee Arthroplasty Using the OrthoPilot and the Software pheno4u TKA Level 1
Brief Title: Study to Evaluate the Performance of Navigated TKA With OrthoPilot® pheno4u TKA Level 1
Acronym: TKA4U
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-25084
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis, Knee; Joint Diseases; Rheumatoid Arthritis of Knee; Posttraumatic Arthropathy
Keywords: Navigation; Total Knee Arthroplasty; OrthoPilot
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pheno4u TKA Level 1: Navigation of TKA (Total Knee Arthroplasty) using the new pheno4uTKA Level 1 software for OrthoPilot Elite®.
  Interventions: Procedure: Navigated Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Navigated Total Knee Arthroplasty — The OrthoPilot® Software Pheno4u TKA Level 1 is an application software for computer aided navigation of surgical instruments and serves (in combination with compatible hardware and compatible navigated instruments) as an optional aid for the surgeon during the preparation of the implant site for a compatible knee endoprosthesis.

SUMMARY:
The purpose of this PMCF study is to demonstrate the accuracy of navigation using the new pheno4uTKA Level 1 software for OrthoPilot Elite® and to evaluate its safety and performance.

Patient-related outcome measures (PROM) will be acquired to investigate functional outcome and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a TKA with the OrthoPilot® Navigation System with a Aesculap total knee endo-prosthesis
* Written signed informed consent of patient
* Willingness and mental ability to participate at the long-term follow-up examinations

Exclusion Criteria:

* Pregnancy
* Patients < 18 years or > 80 years
* Patients unable to participate at the follow-up examination (physically, mentally)
* Previous joint replacement at the index knee
* ASA classification > 3 ( ASA I: A healthy patient without systemic diseases. ASA II: A patient with a mild systemic disease that is well controlled (e.g., well-controlled diabetes or hypertension). ASA III: A patient with a severe systemic disease that causes functional limitations (e.g., poorly controlled diabetes, COPD). ASA IV: A patient with a life-threatening systemic disease (e.g., severe heart failure, sepsis). ASA V: A dying patient who is not expected to survive without the operation. ASA VI: A deceased patient whose organs are being removed for donation.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 80 years of age having indication for a fixed-bearing total knee endoprosthesis, without retropatellar arthrosis requiring patella resurfacing
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the surgical accuracy between the new OrthoPilot Software and the previous OrthoPilot Software | 3 months post OP
  The primary variable delta (aHKA), is defined as the difference in the arithmetic hip-knee-angle (aHKA) between the 3 months postoperative and the intraoperatively planned value. The aHKA is calculated as the difference of the mechanical medial proximal tibial angle (MPTA) and the mechanical lateral distal femoral angle (LDFA), both measured in degrees.

SECONDARY OUTCOMES:
Implant survival | ongoing, up to 2 years follow-up
  Secondary interventions at the index knee
Oxford Knee Score (OKS) | Preoperative,3 months-, 12 months and 2 years post operative
  The Oxford Knee Score (OKS) is a validated joint-specific patient-reported outcome measure that is commonly employed to assess the outcome of TKA. It is a 12-item, patient-reported questionnaire originally developed and validated specifically to assess function and pain in patients undergoing TKA. It is short, reproducible, valid and sensitive to clinically important changes over time. OKS ranges from 0 to 48 with 48 being the best outcome.
Forgotten Joint Score (FJS) | Preoperative,3 months-, 12 months and 2 years post operative
  The FJS-12 contains 12 questions. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score.
  Final score = 100 - ((sum(item01 to item12) - 12)/48*100). Lower scores indicate less awareness of the operated knee during daily activities. The range of the final score is from 0 to 100 (where 0 is worst and 100 means best score)
Quality of Life (EQ-5D-5L) | Preoperative, Postoperative 3 Months + /- 6 weeks, Postoperative 12 months + /- 6 weeks, Postoperative 2 year + /- 3 months
  Quality of life of the patients will be analyzed using the 5-dimensions 5-level measure of the EuroQol Group (EQ-5D-5L), which is a simple and generic measure for clinical and economic assessment.
  The questionnaire covers five different dimensions (mobility, self-care, usual activities,pain/discomfort, anxiety/depression) rated in 5 levels (from "the worst health you can imagine" to "the best health you can imagine"). The questionnaire is filled by the patients themselves.
NET Promotor Score (NPS) | Postoperative 3 Months + /- 6 weeks, Postoperative 12 months + /- 6 weeks, Postoperative 2 year + /- 3 months
  The Net Promoter Score (NPS) was developed for measuring satisfaction in economic research.
  Colloquially, it is referred to as the "friends and family test". In the healthcare sector, the NPS is used as an overarching measure of patient satisfaction. The NPS metric evaluates the likelihood that a patient will recommend the received healthcare service to others. The NPS is assessed using a scale from 1 to 10. A rating between 9 and 10 is classified as a promoter. A rating between 7 and 8 is considered neutral, and a rating between 0 and 6 is deemed a detractor. The overall score is simply calculated by subtracting the percentage of detractors from the percentage of promoters.
  Scores range from -100 (everyone is a detractor) to +100 (everyone is a promoter). In the industry, a positive score is viewed favorably, and scores above 50 are considered indicative of strong performance.
Anterior knee pain | Preoperative,3 months-, 12 months and 2 years post operative
  Anterior knee pain will be used to evaluate the performance of the implantation and the implant itself.
  Rating Description Points:
  0 = No pain (0 Points) I = Mild pain that does not intrude on daily activities (5 Points) II= Moderate pain that is a nuisance; patient not considering further surgery (10 Points) III= Severe pain; patient considering further surgery (15 Points)
Radiological results | Preoperative, Discharge, 1 year post op
  Routinely performed radiographic images are used to evaluate the status of the affected knee, preoperatively, and the status of the implant components, postoperatively. Analysis of parameters will be defined in the radiographic protocol, where precise definition of the implant alignment parameter of the tibial and femoral component by measurement of the LDFA (laterale distale Femurankle) and MPTA (medial proximal Tibiaankle) is given. Both ankles have the same unit and are measured in degrees.
All (Serious) Adverse Events | 2 years
  During the course of the study, any upcoming intra- or postoperative (serious) adverse will be documented. The total number of AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed to assess the safety of the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, Prof. Dr., Principal Investigator — Universitätsklinikum Carl Gustav Carus
Locations (4):
- Šumperk Hospital Inc., Šumperk, Czechia
- Germany (3):
  - Klinikum Konstanz GmbH, Konstanz, Baden-Wurttemberg
  - Park-Klinik Weißensee, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden